CLINICAL TRIAL: NCT06498245
Title: Early Abdominal Wall Prosthesis Infections: Epidemiology, Risk Factors and Factors Linked to Recovery
Acronym: AWPI
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9063
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Wall Prosthesis Infections
Keywords: Abdominal wall prosthesis; Antibiotic therapy; Surgical revision; Abdominal wall

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Abdominal wall prosthesis infections are among the complications most feared by digestive surgeons. Indeed, this complication is associated with high morbidity and is difficult to manage (antibiotic therapy? surgical revision?). Much data is missing in the literature because there are many types of prosthesis, implemented in patients with very varied conditions and the treatment is not strictly speaking codified.

The investigators wish to carry out a retrospective study on approximately 500 patients and research the main characteristics of the different infections (which microorganism? which site? what time of appearance), the factors linked to the appearance of these infections and above all how to optimize their management. charge.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject operated on at the HUS in the department of Pr. Rohr between January 1, 2017 and July 26, 2023
* Operation of an incisional hernia cure with installation of an abdominal wall prosthesis
* Absence of written opposition in the subject's medical file to the reuse of their data for scientific research purposes.

Exclusion Criteria:

* Subject having expressed his opposition to the reuse of his data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) operated on at the HUS in the department of Pr. Rohr between January 1, 2017 and July 26, 2023
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Recovery of wall prosthesis infection after 3 months from the start of the infection | 3 months from the start of the infection of the prothesis

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France